CLINICAL TRIAL: NCT02358135
Title: Collaborative Connected Health (CCH): A Pragmatic Trial Evaluating Effectiveness of CCH in Psoriasis Management Compared to In-person Visits.
Brief Title: Collaborative Connected Health (CCH) for PCORI
Acronym: PCORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, April Armstrong, Associate Dean, Clinical Research, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-15-00417
Record Dates: First submitted 2015-01-06; First posted 2015-02-06 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
Keywords: Pragmatic; Equivalency; Teledermatology
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): In-person care is the control group because it is currently considered the standard of care in delivering dermatologic services. The intervention includes regular visits to a physician, and may include such treatments as ointments, steroids or ultraviolet therapy at the discretion of a physician. In-person care is the major healthcare-delivery model for managing chronic skin diseases and a realistic, primary option that patients face. The patients in the in-person arm can seek psoriasis care from primary care practitioners or dermatologists, just as they would in the real world.
  Interventions: Other: Control
- CCH Model (Experimental): The intervention arm will be the collaborative connected health (CCH) model, which purports to increase access to specialists and improve outcomes. Specifically, CCH offers multiple modalities for patients and primary care providers (PCPs) to access dermatologists online directly and asynchronously. CCH also fosters team care and patient engagement through active sharing of management plans and multidirectional, informed communication among patients, PCPs, and dermatologists.
  Interventions: Other: Collaborative Connected health, (CCH)

INTERVENTIONS:
Other: Collaborative Connected health, (CCH) — CCH is an asynchronous, secure online platform where patients can upload images of psoriasis lesions and submit assessments. Likewise, practitioners can request and/or initiate dermatology consultations, assume longitudinal care or communicate with patients directly.
  Arms: CCH Model
Other: Control — In-person care is the control group because it is currently considered the standard of care in delivering dermatologic services. The intervention includes regular visits to a physician, and may include such treatments as ointments, steroids or UV therapy at the discretion of a physician. In-person care is the major healthcare-delivery model for managing chronic skin diseases and a realistic, primary option that patients face. The patients in the in-person arm can seek psoriasis care from PCPs or dermatologists, just as they would in the real world.
  Arms: Control

SUMMARY:
The investigators propose to evaluate whether an innovative collaborative connected health (CCH) model increases access to specialists and improves patient outcomes. CCH offers multiple modalities for patients and primary care providers (PCPs) to access dermatologists online directly and asynchronously to maximize effectiveness in a real-world setting. CCH also fosters team care and patient engagement through active sharing of management plans and multidirectional, informed communication among patients, PCPs, and dermatologists. The specific aims of the proposal are to (1) determine whether the CCH model results in equivalent improvements in psoriasis disease severity compared to in-person care, (2) determine whether the CCH model results in equivalent improvements in quality of life and mental health compared to in-person care, and (3) assess whether the CCH model provides better access to care than in-person care.

DETAILED DESCRIPTION:
The investigators propose to conduct a 12-month, pragmatic, randomized controlled trial to evaluate the impact of a collaborative connected health model for psoriasis management compared to inperson care. The pragmatic trial will compare psoriasis severity, quality-of-life, mental health, and access-to-care between the two models. We will enroll 300 psoriasis patients from Colorado and California. In addition to recruiting patients from the general population, we will place a specific emphasis on recruiting psoriasis patients living in rural and underserved communities. We will also recruit from the full disease spectrum of mild, moderate, and severe psoriasis patients. We will use an intention-to-treat approach to analyze outcomes and perform longitudinal data analysis using repeated measures approach to identify potential differences in the trend over time between the two arms. To evaluate the utility of CCH for increasing access from patients' and clinicians' perspective, the study team will conduct key informant interviews and use qualitative analytical techniques with investigator triangulation and member checking to enhance the validity of the conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Be age 18 years and older
* Have physician-diagnosed plaque psoriasis
* Have access to internet and a digital camera or a mobile phone with camera features
* Have a primary care provider or the ability to establish primary care

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD MPH, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of California Davis School of Medicine, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado

REFERENCES:
- [Derived] Armstrong AW, Chambers CJ, Maverakis E, Cheng MY, Dunnick CA, Chren MM, Gelfand JM, Wong DJ, Gibbons BM, Gibbons CM, Torres J, Steel AC, Wang EA, Clark CM, Singh S, Kornmehl HA, Wilken R, Florek AG, Ford AR, Ma C, Ehsani-Chimeh N, Boddu S, Fujita M, Young PM, Rivas-Sanchez C, Cornejo BI, Serna LC, Carlson ER, Lane CJ. Effectiveness of Online vs In-Person Care for Adults With Psoriasis: A Randomized Clinical Trial. JAMA Netw Open. 2018 Oct 5;1(6):e183062. doi: 10.1001/jamanetworkopen.2018.3062. PMID 30646223
- [Derived] Armstrong AW, Ford AR, Chambers CJ, Maverakis E, Dunnick CA, Chren MM, Gelfand JM, Gibbons CM, Gibbons BM, Lane CJ. Online Care Versus In-Person Care for Improving Quality of Life in Psoriasis: A Randomized Controlled Equivalency Trial. J Invest Dermatol. 2019 May;139(5):1037-1044. doi: 10.1016/j.jid.2018.09.039. Epub 2018 Nov 24. PMID 30481495

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Person Model (Control): The control arm is the in-person model. Patients randomized to the in-person arm sought psoriasis care from Primary Care Physicians (PCPs) or dermatologists in person.
- Online Model (Collaborative Connected-Health): The intervention arm is the online, collaborative connected-health model: an asynchronous, secure online platform where patients can upload images of psoriasis lesions and submit assessments. The collaborative connected-health model was designed such that any specialist services that usually occur in person could be delivered through asynchronous online healthcare in a flexible and prompt manner. In this pragmatic trial, the PCPs could access the dermatologists online asynchronously via consultation or requesting a dermatologist to assume care of a patient's psoriasis.
  Patients randomized to the online group had the option of accessing dermatologists online asynchronously. During an online visit, the patient would upload clinical images and history and transmit the information to the dermatologist. Using the telehealth platform, the dermatologist would review the transmitted information, make treatment recommendations, prescribe medications, and provide educational materials
Period: Overall Study
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Started | 150 | 150
Randomized | 148 | 148
Completed | 135 | 131
Not Completed | 15 | 19

BASELINE CHARACTERISTICS:
Population: A total of 300 patients were enrolled, and a total of 148 patients each were randomized to the online or in-person groups. All randomized participants received the intended intervention, and all were analyzed for the primary outcome and secondary outcomes. Each participant was followed for 12 months. The analyses were based on intention-to-treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health) | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (14.0) | 49.7 (13.6) | 49.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 74 | 75 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 46 | 100
  Not Hispanic or Latino | 94 | 102 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 6 | 13 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 3 | 5 | 8
  White | 97 | 90 | 187
  More than one race | 36 | 34 | 70
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 148 | 148 | 292
Alcohol Use [Count of Participants; unit: Participants]
  Never | 33 | 36 | 69
  Former | 29 | 38 | 67
  Current | 83 | 69 | 152
  Unknown or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Self-Administered Psoriasis Area and Severity Index (SA-PASI)
Description: Participants are asked to complete self-administered Psoriasis Area and Severity Index (SA-PASI). SA-PASI combines the assessment of lesion severity (erythema, induration, and scale) and the affected areas into a single score between 0 (no disease) to 72 (maximal disease). The primary outcome of the study was the mean percent improvement in SA-PASI averaged over three, six, nine, and 12 months. The percent improvement in SA-PASI was defined as the difference in SA-PASI scores between the baseline and each of the follow-up visits divided by the SA-PASI score from the baseline visit.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Score on a Scale | -0.82 (3.43) | -1.37 (3.33)

2. Secondary Outcome: Improvement in Quality of Life as Measured by Dermatology-Specific, Quality of Life Instruments
Description: Quality of life will be assessed using dermatology-specific, quality of life instruments, Skindex-16 and Dermatology Life Quality Index (DLQI). Scores for these assessments will be compared between patients randomized to the CCH model and in-person care.
  Skindex-16 is a validated and reliable instrument that comprehensively captures the effects of skin disease on health-related quality of life. It discriminates among patients with different effects and is responsive to clinical changes over time. Skindex-16 scores range from 0 (no effect) to 100 (effect experienced all the time), and the responses are aggregated in symptoms, emotions, and functioning subscales.
  The Dermatology Life Quality Index (DLQI) is another validated dermatology-specific quality-of-life instrument that has been used in many psoriasis trials. DLQI scores range from 0 to 30, with higher scores indicating more severe impact on quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Score on a Scale
  Skindex-16 | -2.63 (7.32) | -1.79 (5.92)
  DLQI | -1.18 (4.77) | -1.64 (4.34)

3. Secondary Outcome: Access to Care: Distance Traveled
Description: Access to care is an overall term to capture the transportation to care factors including total distance traveled to see a provider (round-trip driving distance from patient's home to provider's office multiplied by the number of in-person visits during the study period).
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: Kilometers
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Kilometers | 178.8 (577.4) | 2.2 (14.2)

4. Secondary Outcome: Depression Severity
Description: Participants will be assessed for depression severity using the Patient Health Questionnaire (PHQ), a validated, self-administered diagnostic instrument for common mental disorders. The PHQ-9 score can range from 0 to 27 with 0 = "No" depression and 27 = "Severe" depression.
  The PHQ is a validated, self-administered version of the Primary Care Evaluation of Mental Disorders (PRIME-MD) diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) depression criteria as "0" (not at all) to "3" (nearly every day). A PHQ-9 score of 10 or greater has 89% sensitivity and 88% specificity for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively. PHQ-9 is a validated tool for diagnosis of depression and monitoring response to interventions.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Score on a scale | -0.76 (4.66) | -0.4 (3.94)

5. Secondary Outcome: Other Psoriasis Disease Severity Measures
Description: Body surface area (BSA) involvement and patient global assessment (PtGA) will be compared between the patients randomized to the CCH model and the in-person care.
  The BSA assessment is a well-established, validated measure used by psoriasis patients to report percent body surface affected by psoriasis in numerous prior studies. BSA ranges from 0% (no involvement) to 100% (complete body surface affected). The PtGA is a validated instrument that measures the overall psoriasis severity from the patients' perspective.40 PtGA is an ordinal six-point scale ranging from 0 (clear) to 5 (severe).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Score on a scale
  BSA | -1.55 (8.87) | -3.38 (11.08)
  PtGA | -.22 (1.26) | -.37 (1.00)

6. Secondary Outcome: Access to Care: Wait Time
Description: Access to care is an overall term to capture transportation factors including time taken to be seen by a provider. me. Wait time is measured by calculating roundtrip transportation time plus in-office waiting time multiplied by the number of in-person visits during the study period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
Number analyzed (Participants) | 148 | 148
Hours | 4.0 (4.5) | 0.1 (0.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | In-Person Model (Control) | Online Model (Collaborative Connected-Health)
All-Cause Mortality (participants affected / at risk) | 1/148 | 1/148
Serious Adverse Events (participants affected / at risk) | 15/148 | 12/148
Other Adverse Events (participants affected / at risk) | 51/148 | 42/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Model (Control) (N=148) | Online Model (Collaborative Connected-Health) (N=148)
Serious Adverse Event (General disorders) | 2 (2) | 2 (2) — Internal malignancies (excluding skin cancer)
Serious Adverse Event (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) — Exacerbation of Arthritis
Serious Adverse Event (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) — Non-melanoma skin cancers
Serious Adverse Event (Surgical and medical procedures) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Model (Control) (N=148) | Online Model (Collaborative Connected-Health) (N=148)
General adverse event (General disorders) | 51 (51) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02358135/Prot_SAP_000.pdf